CLINICAL TRIAL: NCT02759640
Title: First-in-Human, Dose-Escalation Trial of C-Met Kinase Inhibitor HS-10241 in Subjects With Advanced Solid Tumors
Brief Title: A Phase I Trial of HS-10241 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10241-001
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2019-02

CONDITIONS: Neoplasm; Solid Tumors
Keywords: c-Met kinase inhibitor; Advanced solid tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HS-10241 (Experimental): HS-10241 is administered orally starting at 100 mg/day.
  Interventions: Drug: HS-10241

INTERVENTIONS:
Drug: HS-10241 — HS-10241 is administered orally starting at 100 mg/day.

SUMMARY:
This is a phase 1, open-label, dose-escalation trial of HS-10241 as monotherapy in subjects with solid tumors. HS-10241 will be administered orally once daily.

DETAILED DESCRIPTION:
Recently, c-Met has become an important target of intensive research in search of specific inhibitors as potential new therapies for cancers driven by c-Met activation. HS-10241 is a potent and selective small molecule c-Met kinase inhibitor for both enzyme and c-Met phosphorylation in the cell. Consistent with its potent enzyme and cell activity, HS-10241 was found to inhibit cell growth in vitro against tumors with c-Met gene amplification or c-Met overexpression. On the basis of these findings, the current trial will be conducted in participants with advanced solid tumors for whom standard treatment is not currently available.

This study consists of 2 phases. In the dose-escalation phase, up to 5 dose levels of HS-10241 (100 mg/day, 200 mg/day, 340 mg/day, 500 mg/day, and 700 mg/day) will be investigated with a sequential "3+3" design (3 or 6 participants in every dose level). Participants will have a single-dose pharmacokinetic (PK) run-in period (7 days). Following the first dose, participants will enter a 1 week treatment-free period to evaluate safety and single-dose PK. If no dose-limiting toxicities (DLTs) are observed during the 1-week period, HS-10241 administration will resume at the same dose level.

In the expansion phase, up to 12 additional participants will be enrolled at the MTD. Anti-tumor effects will be assessed every 2 cycles (4 weeks=1 cycle) by using RECIST version 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Ability to understand the purposes and risks of the trial and his/her informed consent using the Human Research Ethics Committee (HREC) approved informed consent form (ICF).
3. Histologically or cytologically confirmed advanced or metastatic solid tumor for which standard therapy does not exist, has failed, or has been refused.
4. Recovered from toxicities of prior anti-cancer treatment to Grade 1 or less (except alopecia)
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Life expectancy of at least 3 months
7. Acceptable liver function defined below:

   * Total bilirubin ≤ 2 times upper limit of normal range (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 times ULN; however, ≤5 times ULN in a subject who has liver metastases
8. Acceptable renal function defined below:

   * Serum creatinine ≤1.5 times ULN or calculated creatinine clearance (by the Cockcroft-Gault formula) ≥60 mL/minutes
9. Acceptable coagulation status defined below:

   * Prothrombin time <1.5 times ULN
   * Partial thrombin time <1.5 times ULN
10. Acceptable hematologic status (without hematologic supports including hematopoietic factor, blood transfusion) defined below:

    * Absolute neutrophil count (ANC) ≥1500/μL
    * Platelet count ≥100000/μL
    * Hemoglobin ≥9.0 g/dL
11. No clinically significant abnormalities in urinalysis
12. All participants must agree to use effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an intrauterine device) with their partner from entry into the trial through 6 months after the last dose.

Exclusion Criteria:

1. Hematologic malignancies
2. Cardiac disease with New York Heart Association (NYHA) Class III or IV, including congestive heart failure, myocardial infarction within 6 months prior to the trial entry, unstable arrhythmia, or symptomatic peripheral arterial vascular disease
3. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
4. Major surgery, other than diagnostic surgery, within 4 weeks prior to the trial entry, without complete recovery
5. Percutaneous coronary intervention conducted within 6 months prior to the trial entry for cardiac infarction or angina pectoris
6. Seizure disorders requiring anticonvulsant therapy
7. Taking a medication that prolongs QT interval and has a risk of Torsade de Pointes, or a history of long QT syndrome
8. Medical history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product
9. Anti-cancer treatment with radiation therapy, surgery, chemotherapy, targeted therapies (erlotinib, lapatinib, etc.), or immunotherapy within 4 weeks (6 weeks for nitrosoureas or Mitomycin C) prior to trial entry. Ongoing androgen deprivation therapy or bisphosphonates are allowed.
10. Participation in an investigational drug or device trial within 4 weeks prior to the trial entry
11. Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
12. Recent venous thrombosis (including deep vein thrombosis or pulmonary embolism within 1 year of trial entry)
13. History of upper gastrointestinal hemorrhage, peptic ulcer disease, or bleeding diathesis;
14. Subject is pregnant (positive serum beta human chorionic gonadotropin [β-HCG] test at Screening) or is currently breast-feeding, their partner anticipates becoming pregnant/impregnating during the trial or within 6 months after receiving the last dose of trial treatment
15. Concomitant disease or condition that could interfere with the conduct of the trial, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this trial
16. History of organ allograft, autologous stem cell transplantation, or allogeneic stem cell transplantation
17. Unwillingness or inability to comply with the trial protocol for any reason
18. Legal incapacity or limited legal capacity
19. Known drug abuse or alcohol abuse
20. Taking a medication that is a moderate or strong inhibitor or inducer of CYP2C9. Patients are eligible if these medications can be stopped or substituted within the screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 4 weeks
  MTD is defined as the maximum dose level at which no more than 1 out of 3 participants experience a DLT within the first 4 weeks of multiple dosing.

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | 24 months
Peak plasma concentration (Cmax) | 4 weeks
Area under the plasma concentration-time curve (AUC） | 4 weeks
T1/2 (half-life) | 4 weeks
Objective response rate (ORR) | 24 months
Time to reach maximum plasma concentration (Tmax) | 4 weeks
Clearance (CL) | 4 weeks
Volume of distribution at steady state (Vss) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Liverpool, Liverpool, New South Wales

IPD SHARING:
Plan to Share IPD: No